CLINICAL TRIAL: NCT04148612
Title: Study to Evaluate the Benefit of the Opti-Me Application to Inform SSRIs, SNRIs Medication Prescription or TMS Treatment for Subjects With a Primary Diagnosis of Major Depression Disorder (MDD)
Brief Title: A Study to Evaluate the Benefit of Opti-Me Application to Different Treatments of MDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ELM-56
Record Dates: First submitted 2019-10-29; First posted 2019-11-01 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opti-Me (Experimental): Patients in this group will be treated based on the Opti-Me algorithm recommended treatment.
  Interventions: Diagnostic Test: Opti-Me
- Randomization (No Intervention): Patients in this group will be treated by random assignment of treatment.

INTERVENTIONS:
Diagnostic Test: Opti-Me — Opti-Me algorithm provides the likelihood of response to the 3 treatment options: SSRIs, SNRIs or TMS in MDD patients.
  Arms: Opti-Me

SUMMARY:
Major depressive disorder (MDD) is a debilitating disease characterized by depressed mood, diminished interests, impaired cognitive function and vegetative symptoms, such as disturbed sleep or appetite. MDD affects one in six adults in their lifetime. To date, decisions regarding specific treatment protocols for MDD are based on clinical experience and risk factors with limited data on outcome prediction. In addition, since it takes 8 weeks to assess if a treatment is successful, the long and often unsuccessful search for an effective antidepressant is accompanied by significant decrease in patients' quality of life, an increased risk of suicidal action, and decreased chance of response and remission with each attempt. This has led to examination of various markers (e.g., neuroimaging, electrophysiological, genetic and behavioral) in an attempt to predict the response to various forms of treatments, including pharmacotherapies and TMS (Transcranial Magnetic Stimulation) for depression.

Elminda had developed a novel, non-invasive imaging EEG-based technology, Brain Network Analytics (BNA), for visualization and quantification of specific brain functions. The rationale of the study is to develop a reliable marker for MDD treatment outcome based on the BNA.

DETAILED DESCRIPTION:
Elminda was granted a specific funding from the European Union in the framework of the Horizon 2020 program (Grant No: 808677 & 859051) to perform this study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with a clinical diagnosis of Major Depressive Disorder (MDD) as defined by the DSM V
2. MDD Patients who in the judgement of their physician require treatment management, and are eligible to receive any of the approved SSRI/SNRI drugs defined in the study protocol or TMS treatment .
3. Males and Females 18-65 years old, inclusive, at the Screening visit.
4. A score of ≥ 20 on the MADRS.
5. History of up to 5 failed MDD pharmacotherapies treatments within the current episode
6. Patients able to understand and sign written informed consent.
7. Patients able and willing to comply with the requirements of the protocol.
8. Female subjects of childbearing potential who are using acceptable birth control measures.

Key Exclusion Criteria:

1. History or presence of epilepsy or seizures or convulsions.
2. History of any progressive neurological disorders in the past five ( 5 ) years.
3. A suicidal attempt within the past year, score 5 on MADRS Item 10 (Suicidal Thoughts) according to investigator judgment based on interview or the C-SSRS questionnaire.
4. Any clinically significant uncontrolled nervous system, gastrointestinal (GI), renal, pulmonary, cardiovascular, or hepatic concomitant disease that in the investigator's opinion would preclude patient participation.
5. Diagnosis of a psychotic disorder.
6. History of or current open head trauma.
7. Metal, shrapnel or other similar objects in the head that could affect the EEG. History of craniotomy, cerebral metastases, cerebrovascular accident;
8. Current diagnosis of schizophrenia, schizo affective disorder, dementia, mental retardation, or major depression with psychotic features;
9. Chronic or acute pain requiring prescription pain medication(s) (narcotic or synthetic narcotic).
10. Participation in any other therapeutic drug study within 60 days preceding inclusion.
11. Deafness, and/or blindness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population will consist of at least 40% Male and 40% Female patients
Enrollment: 390 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The response to treatment based on the Montgomery-Asberg Depression Rating Scale (MADRS) defined as a decline of at least 50% in the MADRS score from Baseline (BL) to the end of treatment (EOT) period which will be defined per treatment type. | up to 8 weeks
Accuracy of the model will be assessed by the specificity and sensitivity of the model developed based on Cohort 1(GR1) and implemented in Cohort 2 Arm A (GR2A). | end of study, estimated 2 years
Comparison of the proportion of responders in Cohort 2 Arm A (GR2A) (assignment to treatment with the guidance of the Opti-Me algorithm) vs Cohort 1 (GR1) + Cohort 2 Arm B (GR2B) (random allocation to treatment). | up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Beer Ya'aqov, Be’er Ya‘aqov, Israel
- University of Zurich Hospital, Zurich, Switzerland